CLINICAL TRIAL: NCT05327140
Title: Reliability of Inflammatory Back Pain Criteria and Activity Scores in Patients With Axial Spondyloarthritis
Brief Title: Reliability of IBP Criteria & Activity Scores in Patients With AxSpA
Acronym: IBP/AxSpA
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Noha Ehab Hamed, Physician, Zagazig University
Other Study IDs: ZU-IRB #6983/13-6-2021
Record Dates: First submitted 2021-12-22; First posted 2022-04-14 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Axial Spondyloarthritis; Inflammatory Back Pain
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with axial spondyloarthritis: ASAS classification criteria which relies either on sacroiliitis on imaging plus one SpA feature (imaging arm) or HLA-B27 antigen plus two SpA features (clinical arm), in a patient with chronic back pain and age at onset of less than 45 years
- patients with mechanical back pain: Patients diagnosed as chronic (more than 3 months) mechanical back pain, the diagnosis has been made prior to the study by the treating specialist, these patients are herein as a control group

SUMMARY:
The current ASAS classification of AxSpA relies either on sacroiliitis on imaging plus one SpA feature (imaging arm) or HLA-B27 antigen plus two SpA features (clinical arm), in a patient with chronic back pain and age at onset of less than 45 years. IBP which is a major symptom of SpA depends more on patient's perception which is not usually accurate. As well, disease activity is measured by ASDAS, BASDAI, and BASFAI which depend more on subjective measures. Assessment of reliability of IBP criteria, ASDAS, BASDAI, and BASFAI in diagnosis and evaluation of activity of AxSpA is essential for better health care.

DETAILED DESCRIPTION:
Axial spondyloarthritis (AxSpA) is a chronic inflammatory disease that affects the axial skeleton mainly leading to significant pain and disability. Early diagnosis of AxSpA is important for better management of symptoms and to limit spinal damage. The last classification of AxSpA is ASAS classification criteria which relies either on sacroiliitis on imaging plus one SpA feature (imaging arm) or HLA-B27 antigen plus two SpA features (clinical arm), in a patient with chronic back pain and age at onset of less than 45 years. Inflammatory back pain (IBP) is the key clinical symptom of AxSpA and is often present at disease onset. There are different sets of IBP criteria which include the Calin criteria , Berlin criteria, and the Assessment of SpondyloArthritis international Society (ASAS) IBP experts criteria. These sets when assessed by different rheumatologists had different sensitivity and specificity.

As IBP has certain characters, taking the clinical history has been considered as a screening test for patients with chronic back pain to identify patients with AxSpA. But, the value of this screening test has been questioned. Disease activity in AxSpA has been measured by the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). It has been used extensively since 1994 but with some limitations as it does not include the physician's assessment of the disease and does not assess the impact of specific clinical factors.

The Bath Ankylosing Spondylitis Functional Index (BASFI) has been also developed as an approach to defining and monitoring functional ability in patients with AxSpA. ASAS developed a disease activity score for patient with AxSpA which is called Ankylosing Spondylitis Disease Activity Score (ASDAS) that combines patient-reported assessments with acute phase reactants (C-reactive protein [CRP] or erythrocyte sedimentation rate [ESR]). However, it is based largely on subjective measures, and lacks objective biomarker of disease activity.

The evaluation of disease activity in AxSpA is complex and multifactorial. Also, patients and physicians have different perspectives of the disease and none of the current single-item or combined indexes adequately unifies both perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Group 1
* Patients diagnosed as AxSpA.
* Age > 18 years and < 45 years at onset of the disease. Group 2
* Patients diagnosed as chronic mechanical back pain.
* Age > 18 years and < 45 years at onset of the disease.

Exclusion Criteria:

* Patients having acute or subacute back pain.
* Patients having back pain referred from another site.
* Patients with any other autoimmune disease: rheumatoid arthritis, systemic lupus erythematosus, Behçet's disease… etc.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Group 1 Patients diagnosed as AxSpA according to the ASAS classification criteria for AxSpA. Group 2 Patients diagnosed as chronic (more than 3 months) mechanical back pain, the diagnosis has been made prior to the study by the treating specialist, these patients are herein as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
assessment of reliability, sensitivity, and specificity of inflammatory back pain criteria (the Assessment of SpondyloArthritis international Society IBP experts criteria) depending on a gold standard which is the global evaluation of the rheumatologist. | 8/2021 to 5/2022
  Assessment of reliability of each item and the whole set of inflammatory back pain criteria ( the Assessment of SpondyloArthritis international Society (ASAS) IBP experts criteria) depending on a gold standard which is the global evaluation of expert rheumatologist: is it inflammatory or mechanical back pain.
  The Assessment of SpondyloArthritis international Society (ASAS) IBP experts criteria includes 5 items: age at onset ≤ 40 years, insidious onset, improvement with exercise, no improvement with rest, pain at night. This set of criteria is achieved if at least four parameters are met.
assessment of reliability of Ankylosing Spondylitis Disease Activity Score in axial spondyloarthritis patients. | 8/2021 to 5/2022
  Ankylosing Spondylitis Disease Activity Score (ASDAS-CRP) includes 4 questions about disease activity (Axial pain, Peripheral Pain/Swelling, Duration of Morning Stiffness, activity of the disease on average during the last week) and CRP. Each question has a score from 0 to 10. 0 means no, and 10 means sever.
  ASDAS_CRP = 0.121 × total back pain + 0.110 × patient global + 0.073 × peripheral pain / swelling + 0.058 × duration of morning stiffness + 0.579 × Ln (CRP+1).
  ASDAS scores : <1.3 "inactive disease" and <2.1"low disease activity", ≤3.5 "high disease activity", and >3.5 "very high disease activity".
  The score is applied to the same group of patients by 2 rheumatologists. The scores of each question and the total score that detected by the two rheumatologists are compared to detect agreement between the two rheumatologist and assess reliability of this score

CONTACTS AND LOCATIONS:
Overall Officials: Eman El-shahawy, Study Director — Zagazig University; Mohamed Mortada, Study Director — Zagazig University; Safaa Elnaggar, Study Director — Zagazig University; Noha Hamed, Principal Investigator — Zagazig University
Locations (1):
- Zagazig university, Zagazig, Sharqia Province, Egypt

REFERENCES:
- [Background] Calin A, Porta J, Fries JF, Schurman DJ. Clinical history as a screening test for ankylosing spondylitis. JAMA. 1977 Jun 13;237(24):2613-4. PMID 140252
- [Background] Calin A, Garrett S, Whitelock H, Kennedy LG, O'Hea J, Mallorie P, Jenkinson T. A new approach to defining functional ability in ankylosing spondylitis: the development of the Bath Ankylosing Spondylitis Functional Index. J Rheumatol. 1994 Dec;21(12):2281-5. PMID 7699629
- [Background] Deodhar A, Blanco R, Dokoupilova E, Hall S, Kameda H, Kivitz AJ, Poddubnyy D, van de Sande M, Wiksten AS, Porter BO, Richards HB, Haemmerle S, Braun J. Improvement of Signs and Symptoms of Nonradiographic Axial Spondyloarthritis in Patients Treated With Secukinumab: Primary Results of a Randomized, Placebo-Controlled Phase III Study. Arthritis Rheumatol. 2021 Jan;73(1):110-120. doi: 10.1002/art.41477. Epub 2020 Nov 24. PMID 32770640
- [Background] Garrett S, Jenkinson T, Kennedy LG, Whitelock H, Gaisford P, Calin A. A new approach to defining disease status in ankylosing spondylitis: the Bath Ankylosing Spondylitis Disease Activity Index. J Rheumatol. 1994 Dec;21(12):2286-91. PMID 7699630
- [Background] Machado P, van der Heijde D. How to measure disease activity in axial spondyloarthritis? Curr Opin Rheumatol. 2011 Jul;23(4):339-45. doi: 10.1097/BOR.0b013e3283470f23. PMID 21519269
- [Background] Poddubnyy D, Callhoff J, Spiller I, Listing J, Braun J, Sieper J, Rudwaleit M. Diagnostic accuracy of inflammatory back pain for axial spondyloarthritis in rheumatological care. RMD Open. 2018 Dec 5;4(2):e000825. doi: 10.1136/rmdopen-2018-000825. eCollection 2018. PMID 30713715
- [Background] Reveille JD. Biomarkers for diagnosis, monitoring of progression, and treatment responses in ankylosing spondylitis and axial spondyloarthritis. Clin Rheumatol. 2015 Jun;34(6):1009-18. doi: 10.1007/s10067-015-2949-3. Epub 2015 May 5. PMID 25939520
- [Background] Ritchlin C, Adamopoulos IE. Axial spondyloarthritis: new advances in diagnosis and management. BMJ. 2021 Jan 4;372:m4447. doi: 10.1136/bmj.m4447. PMID 33397652
- [Background] Rudwaleit M, Metter A, Listing J, Sieper J, Braun J. Inflammatory back pain in ankylosing spondylitis: a reassessment of the clinical history for application as classification and diagnostic criteria. Arthritis Rheum. 2006 Feb;54(2):569-78. doi: 10.1002/art.21619. PMID 16447233
- [Background] Rudwaleit M, Landewe R, van der Heijde D, Listing J, Brandt J, Braun J, Burgos-Vargas R, Collantes-Estevez E, Davis J, Dijkmans B, Dougados M, Emery P, van der Horst-Bruinsma IE, Inman R, Khan MA, Leirisalo-Repo M, van der Linden S, Maksymowych WP, Mielants H, Olivieri I, Sturrock R, de Vlam K, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part I): classification of paper patients by expert opinion including uncertainty appraisal. Ann Rheum Dis. 2009 Jun;68(6):770-6. doi: 10.1136/ard.2009.108217. Epub 2009 Mar 17. PMID 19297345
- [Background] Sieper J, van der Heijde D, Landewe R, Brandt J, Burgos-Vagas R, Collantes-Estevez E, Dijkmans B, Dougados M, Khan MA, Leirisalo-Repo M, van der Linden S, Maksymowych WP, Mielants H, Olivieri I, Rudwaleit M. New criteria for inflammatory back pain in patients with chronic back pain: a real patient exercise by experts from the Assessment of SpondyloArthritis international Society (ASAS). Ann Rheum Dis. 2009 Jun;68(6):784-8. doi: 10.1136/ard.2008.101501. Epub 2009 Jan 15. PMID 19147614
- [Background] van der Heijde D, Lie E, Kvien TK, Sieper J, Van den Bosch F, Listing J, Braun J, Landewe R; Assessment of SpondyloArthritis international Society (ASAS). ASDAS, a highly discriminatory ASAS-endorsed disease activity score in patients with ankylosing spondylitis. Ann Rheum Dis. 2009 Dec;68(12):1811-8. doi: 10.1136/ard.2008.100826. Epub 2008 Dec 5. PMID 19060001